CLINICAL TRIAL: NCT00437905
Title: Balloon Angioplasty vs. Cutting Balloon Angioplasty of Femoropopliteal Arteries- a Randomized Controlled Trial
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Version 2.0-12/2003
Record Dates: First submitted 2007-02-20; First posted 2007-02-21 (Estimated); Last update posted 2007-02-21 (Estimated); Status verified 2007-02

CONDITIONS: Peripheral Vascular Disease; Intermittent Claudication; Atherosclerosis; Angioplasty
Keywords: peripheral vascular disease; percutaneous transluminal angioplasty; cutting balloon; balloon angioplasty; randomized controlled trial; restenosis; inflammation
MeSH Terms: conditions — Peripheral Vascular Diseases; Intermittent Claudication; Atherosclerosis; Inflammation | interventions — Angioplasty

INTERVENTIONS:
Procedure: angioplasty

SUMMARY:
The purpose of this study to compare balloon angioplasty (PTA) vs. cutting balloon angioplasty (CB-PTA) in terms of patency and postintervention inflammation in peripheral artery disease.

DETAILED DESCRIPTION:
Balloon Angioplasty is a minimal invasive technique for treatment of superficial femoropoliteal artery obstructions. Despite high initial success rate and an acceptably low complication rate, long-term-results are disappointing as restenosis may frequently occur. One of the hypothesis for the differences in the reported patency rates is that the amount of vessel trauma correlates directly to the prognosis (restenosis) of the treated vessel wall segment.

With the introduction of cutting balloons the problems of elastic recoil and residual stenosis might be resolved, by reduction of vessel wall trauma, vessel wall inflammation and consequently reduced neointima formation.

The promising results especially in coronary arteries led us to initiate a RCT comparing primary PTA vs. CB-PTA for treatment of femoropoliteal obstructions in patients with intermittent claudication or critical limb ischemia.

ELIGIBILITY:
Inclusion Criteria:

* Severe intermittent claucication (Fontaine stage IIb)or limb ischemia, femoropoliteal stenosis/occlusion up to 5 cm length

Exclusion Criteria:

* Previous bypass surgery at the site of treatment,
* Previous stent placement at or immediatly adjacent to target lesion,
* History of anti-platelet-therapy intolerance or adverse reaction to heparin,
* Bleeding diathesis,
* Creatinine > 2,5 mg/dL,
* Active bacterial infection,
* Allergy to contrast media

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2003-06; Study Completion 2007-01

PRIMARY OUTCOMES:
course of postintervention inflammation as indicated by serum levels of C-reactive Protein (CRP+ us-CRP)

SECONDARY OUTCOMES:
occurence of restenosis within 6 months after endovascular treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jasmin Amighi, MD, Principal Investigator — Medical University of Vienna; Martin Schillinger, MD, Principal Investigator — Medical University of Vienna; Manfred Cejna, MD, Principal Investigator — Medical University of Vienna

REFERENCES:
- [Derived] Amighi J, Schillinger M, Dick P, Schlager O, Sabeti S, Mlekusch W, Haumer M, Mathies R, Heinzle G, Schuster A, Loewe C, Koppensteiner R, Lammer J, Minar E, Cejna M. De novo superficial femoropopliteal artery lesions: peripheral cutting balloon angioplasty and restenosis rates--randomized controlled trial. Radiology. 2008 Apr;247(1):267-72. doi: 10.1148/radiol.2471070749. Epub 2008 Feb 12. PMID 18270378